CLINICAL TRIAL: NCT00455624
Title: Prospective Study of Insulin Resistance and Cardiovascular Disease Risk During Androgen Deprivation Therapy for Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Matthew R. Smith, MD, PhD, Professor of Medicine, Massachusetts General Hospital
Other Study IDs: 02-256
Record Dates: First submitted 2007-04-02; First posted 2007-04-04 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Prostate Cancer
Keywords: androgen deprivation therapy; insulin resistance
MeSH Terms: conditions — Prostatic Neoplasms; Insulin Resistance | interventions — Androgen Antagonists

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Androgen deprivation therapy — According to standard medical care

SUMMARY:
The purpose of this study is to find out if androgen deprivation therapy affects insulin, cardiac risk factors such as cholesterol level, and body fat and muscle.

DETAILED DESCRIPTION:
* This is a non-treatment study. This study has no effect on the care the participant will receive.
* In addition to the participants routine standard medical appointments they will need to make 2 additional outpatient visits for special testing over 12 weeks. These 2 additional outpatient visits will include the following: 1) urine and blood tests, 2) Oral Glucose Tolerance Test (OGTT) 3) Body measurements with a tape measure of your arms, legs, and waist and 4) x-ray evaluations (CT scan and bone density test).

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the prostate, clinical stage M0
* About to initiate GnRH agonist therapy
* Karnofsky Performance Status 90 or 100
* Serum creatinine < 2.0mg/dl

Exclusion Criteria:

* Hormone therapy within 12 months
* History of diabetes mellitus or glucose intolerance
* Anabolic agents or metabolic agents known to affect insulin or glucose levels
* Prior hormone therapy within the past 12 months and planned hormone therapy during the 12 week study (Group 2)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men identified with prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2002-11; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
insulin sensitity | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Smith, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

REFERENCES:
- [Background] Smith MR, Lee H, Nathan DM. Insulin sensitivity during combined androgen blockade for prostate cancer. J Clin Endocrinol Metab. 2006 Apr;91(4):1305-8. doi: 10.1210/jc.2005-2507. Epub 2006 Jan 24. PMID 16434464